CLINICAL TRIAL: NCT00697684
Title: A Reduced Intensity Conditioning With Clofarabine Antithymocyte Globulin and Total Lymphoid Irradiation Followed by Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Reduced Intensity Conditioning With Clofarabine, Antithymocyte Globulin (ATG), Total Lymphoid Irradiation (TLI) Followed by Allogeneic Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, David Avigan, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-384
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Acute Lymphocytic Leukemia; Relapsed/Refractory Chronic Lymphocytic Leukemia; Relapsed/Refractory Non Hodgkin's Lymphoma; Hodgkins Disease; Relapsed Refractory Multiple Myeloma
Keywords: Reduced Intensity Allogeneic Stem Cell Transplant; Clofarabine; Rabbit Antithymocyte Globulin; Total Lymphoid Radiation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma | interventions — Antilymphocyte Serum; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (No Intervention): Transplant conditioning will begin day -11 with 5 days of TLI at a dose of 80 cGy per day administered in conjunction with rabbit ATG at a dose of 1.5 mg/kg per day (day -11 to -7). TLI will be completed at 80 cGy per day (day -4 to 0) for a total of 10 fractions (800 cGy).
- Cohort 2 (Experimental): Transplant conditioning will begin day -11 with 5 days of TLI at a dose of 80 cGy per day administered in conjunction with rabbit ATG at a dose of 1.5 mg/kg per day (day -11 to -7). Clofarabine will be given at 20mg/m2/d IV infused over 1 hour x 5 days (day -6 to -2), for a total dose of 100 mg/m(2). TLI will be completed at 80 cGy per day (day -4 to 0) for a total of 10 fractions (800 cGy).
  Interventions: Drug: Antithymocyte Globulin; Drug: Clofarabine
- Cohort 3 (Experimental): Transplant conditioning will begin day -11 with 5 days of TLI at a dose of 80 cGy per day administered in conjunction with rabbit ATG at a dose of 1.5 mg/kg per day (day -11 to -7). Clofarabine will be given at 30mg/m2/d IV infused over 1 hour x 5 days (day -6 to -2), for a total dose of 150 mg/m(2). TLI will be completed at 80 cGy per day (day -4 to 0) for a total of 10 fractions (800 cGy).
  Interventions: Drug: Antithymocyte Globulin; Drug: Clofarabine
- Cohort 4 (Experimental): Transplant conditioning will begin day -11 with 5 days of TLI at a dose of 80 cGy per day administered in conjunction with rabbit ATG at a dose of 1.5 mg/kg per day (day -11 to -7). Clofarabine will be given at 40mg/m2/d IV infused over 1 hour x 5 days (day -6 to -2), for a total dose of 200 mg/m(2). TLI will be completed at 80 cGy per day (day -4 to 0) for a total of 10 fractions (800 cGy).
  Interventions: Drug: Antithymocyte Globulin; Drug: Clofarabine

INTERVENTIONS:
Drug: Antithymocyte Globulin
  Arms: Cohort 2; Cohort 3; Cohort 4
Drug: Clofarabine — Transplant conditioning will begin day -11 with 5 days of TLI at a dose of 80 cGy per day administered in conjunction with rabbit ATG at a dose of 1.5 mg/kg per day (day -11 to -7). Clofarabine will be given at 20mg/m2/d IV infused over 1 hour x 5 days (day -6 to -2), for a total dose of 100 mg/m(2). TLI will be completed at 80 cGy per day (day -4 to 0) for a total of 10 fractions (800 cGy).
  Arms: Cohort 2; Cohort 3; Cohort 4
Drug: Clofarabine — Transplant conditioning will begin day -11 with 5 days of TLI at a dose of 80 cGy per day administered in conjunction with rabbit ATG at a dose of 1.5 mg/kg per day (day -11 to -7). Clofarabine will be given at 30mg/m2/d IV infused over 1 hour x 5 days (day -6 to -2), for a total dose of 150 mg/m(2). TLI will be completed at 80 cGy per day (day -4 to 0) for a total of 10 fractions (800 cGy).
  Arms: Cohort 2; Cohort 3; Cohort 4
Drug: Clofarabine — Transplant conditioning will begin day -11 with 5 days of TLI at a dose of 80 cGy per day administered in conjunction with rabbit ATG at a dose of 1.5 mg/kg per day (day -11 to -7). Clofarabine will be given at 40mg/m2/d IV infused over 1 hour x 5 days (day -6 to -2), for a total dose of 200 mg/m(2). TLI will be completed at 80 cGy per day (day -4 to 0) for a total of 10 fractions (800 cGy).
  Arms: Cohort 2; Cohort 3; Cohort 4

SUMMARY:
This study will examine the safety of clofarabine, TLI and ATG as a reduced conditioning regimen prior to allogeneic transplantation. The impact of the conditioning regimen on the presence of the circulating regulatory as compared to activated T cell populations will be assessed.The recovery of DC populations post-transplant will be examined, along with the effect of the regimen on disease free and overall survival.

DETAILED DESCRIPTION:
One approach to limit the toxicity of allogeneic transplantation has been the use of nonmyeloablative regimens preceding the infusion of allogeneic cells.In this strategy, patients receive immunosuppressive therapy that allows for the engraftment of donor cells without the immediate eradication of patient hematopoiesis.The primary mechanism by which the underlying disease is eradicated is not through chemotherapy mediated cytoreduction, but rather through the donor lymphocyte mediated graft versus tumor effect.As a result, patients experience far less regimen related toxicity.Therefore, the adoption of this strategy may allow for the use of allogeneic transplantation in disease settings and patient populations for which it had not been readily applicable in the past.

Over the past several years, the use nonmyeloablative transplant has rapidly expanded.Several reduced intensity conditioning regimens have been developed including fludarabine and cyclophosphamide; fludarabine and melphalan; fludarabine, ATG and low dose busulfan; and fludarabine and low dose TBI. Investigators have demonstrated the feasibility of this treatment approach with the majority of patients demonstrating donor engraftment,decreased regimen related toxicity, and graft mediated regression of disease.In some studies, patients demonstrate a period of mixed donor/host chimerism in which the infusion of donor lymphocytes is associated with achievement of complete donor chimerism.

Although regimen related toxicity is decreased following reduced intensive conditioning regimens, graft versus host disease and opportunistic infections remain a significant source of morbidity and mortality following nonmyeloablative allogeneic transplantation. The impact of nonmyeloablative transplantation on immunological reconstitution has not been fully defined. Persistence of host antigen presenting cells in the post-transplant period may increase the incidence of GVHD due to the presentation of alloantigens to donor T cells. In contrast, residual host cellular immunity may provide enhanced protection against infectious pathogens and allow for more rapid education of donor lymphocytes.

The use of clofarabine in place of fludarabine in combination with cyclophosphamide may augment the anti-leukemia effect of the regimen, enhance cytoreduction, and increase the efficacy of reduced intensity allogeneic transplantation in this setting.A potential issue associated with the use of clofarabine and cyclophosphamide as pre-transplant conditioning is whether the regimen would be sufficiently immunosuppressive to reliably facilitate engraftment of donor hematopoiesis.Another concern relates to the significant incidence of graft versus host disease which remains a major source of morbidity and mortality following reduced intensity transplantation.The use of TLI and ATG has been studied in the context of allogeneic transplantation and has been shown to effectively support engraftment in animal models and clinical trials.TLI has been shown to promote immune tolerance resulting in a decrease in the incidence of graft versus host disease (GVHD).It has been shown to decrease the incidence of rejection following transplantation of a T cell depleted allograft.The conditioning regimen of TLI and cyclophosphamide results in successful engraftment in patients with aplastic anemia.

Regulatory T cells represent a population of T lymphocytes that demonstrate an immunosuppressive phenotype and play an important role in the prevention of autoimmunity and transplant rejection.Regulatory cells express the inhibitory cytokines IL-10 and TGFβ and are thought to suppress immune activation through direct cell contact.Similar to activated effector cells they coexpress CD4 and CD25.Regulatory T cells may be identified by the high levels of CD25 expression and the presence of CTLA-4 and FOXP3.Regulatory T cells demonstrate minimal proliferation to allogeneic stimuli and inhibit third party mixed lymphocyte responses. Increased presence of regulatory T cells have been found in the tumor bed, draining lymph nodes, and circulation in patients with malignancy and inhibit host anti-tumor immune responses.

There has been increasing interest in evaluating the role of regulatory T cells as a means of inhibiting graft versus host disease. In animal models, selective introduction of regulatory T cells prevents the development of graft versus host disease without compromising immune reconstitution or anti-tumor immunity. A variety of strategies for the ex vivo expansion and isolation of regulatory T cells have been explored. A limiting factor has been the similar patterns of expression of cell surface markers between regulatory and activated T cell populations. iNKT cells represent another population of immunomodulatory cells thought to be essential for the generation of tolerance.In pre-clinical models, TLI has been shown to modulate immune effector cells resulting in increased levels of circulating regulatory T cells, preventing GVHD in a mismatched transplant setting.It is thought that iNKT cells are selectively preserved after TLI which polarize T cells towards an inhibitory phenotype. In a clinical study, 37 patients with lymphoid malignancies or acute leukemia underwent conditioning with TLI administered as 10 fractions of 80cGy and ATG.Only 2 patients developed acute GVHD despite the observation of a graft versus disease effect.Of note, a significant increase in the number of donor CD4+ T cells expressing IL-4 was observed suggesting that the immune modulation resulting from TLI/ATG polarized cells towards a TH-2 phenotype.As such, TLI/ATG would like facilitate engraftment and decrease the incidence of GVHD in patients undergoing conditioning with clofarabine.Most importantly, by modulating the host immune effectors but not depleting donor T cells, this strategy should not significantly inhibit the graft versus tumor effect.The prevalence of dendritic cell (DC) subsets (DC1 vs. DC2) in the hematopoietic graft have also been shown to effect the risk of GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a)acute myeloid leukemia exclusive of patients in first complete remission with good risk cytogenetics (translocation 8,21,translocation 15, 17 or inversion 16); B)myelodysplastic syndrome; c)acute lymphocytic leukemia exclusive of patients in first remission without negative prognostic markers; d) relapsed or refractory nonHodgkin's lymphoma or Hodgkin's disease; e)relapsed or refractory multiple myeloma or f)relapsed or refractory chronic lymphocytic leukemia.
2. Patients who are considered appropriate for reduced intensity transplantation must present with at least one of the following: A. Age over 50 B. History of a prior hematopoietic stem cell transplant C. Patient with compromised organ function or comorbid conditioning such that a standard ablative transplant would be considered high risk. D. Patient with low grade Lymphoma or CLL for which reduced intensity transplant would be the optimal therapy compared to an ablative regimen
3. Patients will have a related or unrelated donor matched at 5/6 or 6/6 HLA loci.
4. Patients must be greater than or equal to 18 years old, and younger than or equal to 75 years old to participate in the study.
5. Patients must have ECOG performance status of 0-2
6. Pulmonary function tests demonstrate DLCO (adjusted for Hgb)>50% predicted
7. Cardiac ejection fraction >40%
8. Laboratories:

   * Bilirubin less than or equal to 1.5mg/dL x ULN
   * AST/ALT/Alkaline Phosphatase less than or equal to 2.5x ULN
   * Serum creatinine less than or equal to 1.0mg/dL; if serum creatinine > 1.0MG/dL, then the estimated glomerular filtration rate (GFR) must be >60mL/min/1.73m^2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GRF (ml/min/1.73m^2)=186x (serum creatinine)^1.154x(age in years)^-0.203x(0.742 if patient is female) x (1.212 if patient is black)
9. Patients with serologic evidence of hepatitis B or C exposure will undergo liver biopsy to assess for presence of active hepatitis or fibrosis and quantification of risk of proceeding with transplant.

10. All patients must be capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent. All patients must be informed of the investigational nature of this study and must give written informed consent in accordance with institutional and federal guidelines.

11. Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.

12. Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment

Exclusion Criteria:

1. Patients who are HIV+ will be excluded.
2. Patients must not have serious intercurrent illness such as uncontrolled systemic infection or significant organ compromise which significantly increases the risk of undergoing allogeneic transplantation.
3. Pregnant and lactating women will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-06; Primary Completion 2020-12 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
To assess the toxicity and donor engraftment following treatment with a reduced intensity preparative regimen consisting of clofarabine, rabbit antithymocyte globulin (ATG), and total lymphoid irradiation followed by the infusion of allogeneic stem cells | 30 days

SECONDARY OUTCOMES:
To determine the incidence of acute and chronic graft versus host disease following clofarabine, rabbit ATG, total lymphoid irradiation, and allogeneic transplantation. | 1 year
2. To evaluate the nature of immunologic reconstitution in patients treated clofarabine, rabbit ATG, total lymphoid irradiation, and allogeneic transplantation. The impact of the regimen on the phenotypic and functional characteristics of dendritic cell | 1 year
To determine the disease free survival and overall survival of patients undergoing allogeneic transplantation following following clofarabine, rabbit ATG, and total lymphoid irradiation. | Patient lifetime

CONTACTS AND LOCATIONS:
Overall Officials: David E Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts